CLINICAL TRIAL: NCT00429481
Title: Study to Assess Efficacy, Immunogenicity, Reactogenicity and Safety of Two Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus Vaccine at Different Viral Concentrations in Healthy Infants Previously Uninfected With Human Rotavirus and Approximately 3 Months of Age.
Brief Title: Assess Efficacy, Immune Response & Safety of 2 Doses of Oral Live Attenuated HRV Vaccine at Different Viral Concentrations in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444563/007
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Oral live attenuated human rotavirus vaccine; Gastroenteritis; Vomiting
MeSH Terms: conditions — Hepatitis B; Gastroenteritis; Vomiting | interventions — RIX4414 vaccine

INTERVENTIONS:
Biological: Rotarix

SUMMARY:
To assess the efficacy, immune response and safety of 2 doses of HRV vaccine (at different concentrations) in healthy infants aged approximately 3 months previously uninfected with human rotavirus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 11 and 17 weeks of age at the time of the first vaccination, born after a normal gestation period (between 36 and 42 weeks).
* Written informed consent obtained from the parents or guardians of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous vaccination against or history of or intercurrent diphtheria, tetanus, pertussis, polio and/or Hib.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. (Topical steroids are allowed.)
* Use of antibiotics during the period starting from 7 days before each dose of vaccine(s) and ending 7 days after.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract or other serious medical condition as determined by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* GE within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Household contact with an immunosuppressed individual or pregnant woman.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* Previous confirmed occurrence of RV GE.

Ages: 11 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2464 (Actual)
Dates: Start 2001-01; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of any RV GE

SECONDARY OUTCOMES:
Occurrence of severe RV GE, rotavirus IgA antibody titres, solicited symptoms (Day 0-15), unsolicited Adverse Events (D0-42), Serious Adverse Events (full study),

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] De Vos B, Vesikari T, Linhares AC, Salinas B, Perez-Schael I, Ruiz-Palacios GM, Guerrero Mde L, Phua KB, Delem A, Hardt K. A rotavirus vaccine for prophylaxis of infants against rotavirus gastroenteritis. Pediatr Infect Dis J. 2004 Oct;23(10 Suppl):S179-82. doi: 10.1097/01.inf.0000142370.16514.4a. PMID 15502699
- [Background] De Vos B, Han HH, Bouckenooghe A, Debrus S, Gillard P, Ward R, Cheuvart B. Live attenuated human rotavirus vaccine, RIX4414, provides clinical protection in infants against rotavirus strains with and without shared G and P genotypes: integrated analysis of randomized controlled trials. Pediatr Infect Dis J. 2009 Apr;28(4):261-6. doi: 10.1097/INF.0b013e3181907177. PMID 19289978
- [Background] Phua KB, Quak SH, Lee BW, Emmanuel SC, Goh P, Han HH, De Vos B, Bock HL. Evaluation of RIX4414, a live, attenuated rotavirus vaccine, in a randomized, double-blind, placebo-controlled phase 2 trial involving 2464 Singaporean infants. J Infect Dis. 2005 Sep 1;192 Suppl 1:S6-S16. doi: 10.1086/431511. PMID 16088807
- [Background] Phua KB, Emmanuel SC, Goh P, Quak SH, Lee BW, Han HH, Ward RL, Bernstein DI, De Vos B, Bock HL. A rotavirus vaccine for infants: the Asian experience. Ann Acad Med Singap. 2006 Jan;35(1):38-44. PMID 16470273
- [Background] Phua KB, Quak SH, Emmanuel S, Goh PS, Han HH, Hardt K, Bock HL, De Vos B. A short report on highlights of worldwide development of RIX4414: a Singaporean experience. Vaccine. 2006 May 1;24(18):3782-3. doi: 10.1016/j.vaccine.2006.03.040. Epub 2006 Mar 23. PMID 16600443
- [Background] Phua KB, Quak SH, Lim FS, Goh P, Teoh YL, Datta SK, Han HH, Bock HL. Immunogenicity, reactogenicity and safety of a diphtheria-tetanus-acellular pertussis-inactivated polio and Haemophilus influenzae type b vaccine in a placebo-controlled rotavirus vaccine study. Ann Acad Med Singap. 2008 Jul;37(7):546-53. PMID 18695765
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 444563/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register